CLINICAL TRIAL: NCT00808678
Title: Comparison of the Bioavailability of Fenofibric Acid and Rosuvastatin From ABT-143 Relative to That From the Coadministration of ABT-335 (Fenofibric Acid) and Rosuvastatin Calcium
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: M10-662
Record Dates: First submitted 2008-12-02; First posted 2008-12-16 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2012-09

CONDITIONS: Healthy
Keywords: Adverse Events
MeSH Terms: interventions — 2-(4-(4-chlorobenzoyl)phenoxy)-2-methylpropanoic acid; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): ABT-143 capsules 20/135 mg
  Interventions: Drug: ABT-143
- 2 (Active Comparator): ABT-335 135 mg and rosuvastatin 20 mg
  Interventions: Drug: ABT-335; Drug: rosuvastatin

INTERVENTIONS:
Drug: ABT-143 — once, see arm description for more information
  Arms: 1
Drug: ABT-335 — once, see arm description for more information
  Arms: 2
Drug: rosuvastatin — once, see arm description for more detail
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the safety and compare the pharmacokinetic parameters from the fixed dose combination ABT-143 relative to that from the co-administration of the two monotherapies.

ELIGIBILITY:
Inclusion Criteria:

1. A condition of general good health
2. BMI 19 to 29

Exclusion Criteria:

1. Currently enrolled in another clinical study
2. Females who are pregnant or breast-feeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2008-12; Primary Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of ABT-143 vs (ABT-335 + rosuvastatin) in healthy adults | 7 days
To determine the pharmacokinetic profile(s) for ABt-143 vs. (ABT-335 + rosuvastatin) in healthy adults | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Torbjörn Lundström, MD, Study Director — AstraZeneca
Locations (1):
- Site Reference ID/Investigator# 14762, Orlando, Florida, United States